CLINICAL TRIAL: NCT01678404
Title: A Phase II Study of 131I-rituximab for Patients With Relapsed or Refractory Marginal Zone B-cell Lymphoma
Brief Title: 131I-rituximab for Relapsed or Refractory Marginal Zone B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZL 131I-rituximab RIT
Record Dates: First submitted 2012-09-04; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Relapsed or Refractory Marginal Zone B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell, Marginal Zone | interventions — 131I-rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131I-rituximab (Experimental): 131I-rituximab treatment interval at least 4 weeks up to maximum 6 cycles
  Interventions: Drug: 131I-rituximab

INTERVENTIONS:
Drug: 131I-rituximab

SUMMARY:
Marginal zone B-cell lymphoma (MZL) is a lymphoma originated from B-cell in lymph node with variable differentiation status, which is distributed to a variety of organs.

A high response rate and long term survival is possible through surgery or radiation therapy alone in the case of limited disease. However frequent relapse and progression is observed despite of long term survival. The treatment after relapse has not been established yet.

So we investigate the efficacy of radioimmunotherapy using 131I-rituximab in refractory or relapsed patients with MZL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed marginal zone B-cell lymphoma
* relapsed or refractory patients after treatment including chemotherapy, radiation therapy, and surgery
* Eastern Cooperative Oncology Group performance status ≤ 2
* age≥ 20 years
* More than one measurable lesion (More than 2cm sized lesion in conventional CT scan, More than 1cm sized lesion in spiral CT or contrast-enhanced PET/CT )
* Adequate renal function (serum creatinine ≤ 2.0 mg/dl or Ccr ≥ 60 ml/min)
* Adequate hepatic function (serum bilirubin ≤ 2.0 mg/dl , AST/ALT ≤ 3 upper normal limit)
* Adequate bone marrow reservoir (ANC ≥1,500/㎕, platelet count≥ 75,000/㎕)
* patient who agree the purpose and intention of this clinical trial

Exclusion Criteria:

* recent (<5 years) history of other malignancy or unrecovered from the disease (appropriately treated skin cancer and uterine cervix carcinoma in situ are excluded)
* hemodynamically unstable due to the recent (<12 months) history of severe heart disease such as myocardial infarction
* acute complications of severe lung or metabolic disease
* Combined severe neurological or psychiatric disease
* Unrecovered from infection or other medical disease
* Recent (<30 days) history of enrollment of other clinical trial
* Pregnant or breast-feeding woman
* women of childbearing potential and men not employing adequate contraception at least for 1 year
* Previous history drug allergy to the content of 131I-rituximab
* Infection(sepsis, pneumonia, viral infection, etc) (inactivated hepatitis B carrier can be enrolled)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 5 years
  International Working Group Response criteria

SECONDARY OUTCOMES:
Response duration | up to 5 years
Progression free survival | up to 5 years
Overall survival | up to 5 years
Number of Adverse Events | up to 5 years
  grading the adverse events using CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Kang, M.D., Principal Investigator — Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences
Locations (1):
- Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences, Seoul, South Korea